CLINICAL TRIAL: NCT05910125
Title: Aspirin Combined With Clopidogrel Versus Intravenous Alteplase for Acute Minor Stroke: An Open-label, Blinded Endpoint, Randomized Controlled Trial
Brief Title: Aspirin Combined With Clopidogrel Versus Intravenous Alteplase for Acute Minor Stroke
Acronym: AGREE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2022-252-02
Record Dates: First submitted 2023-06-11; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Clopidogrel; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAPT group (Experimental): Receiving dual antiplatelet therapy immediately after randomization (Oral aspirin 100mg+clopidogrel 300mg, Day 1). Participants who show no evidence of intracranial hemorrhage on skull CT 24 hours after randomization will receive oral aspirin 100mg/d (Day 2-90) and clopidogrel 75mg/d (Day 2-21), while those with intracranial hemorrhage on skull CT will not receive any antiplatelet drugs.
  Interventions: Drug: Aspirin; Drug: Clopidogrel
- IVT group (Active Comparator): Receiving intravenous thrombolysis immediately after randomization (Intravenous alteplase, 0.9mg/kg, a maximum dosage of 90mg). Participants who show no evidence of intracranial hemorrhage on skull CT 24 hours after randomization will receive oral aspirin 100mg/d (Day 2-90), while those with intracranial hemorrhage on skull CT will not receive any antiplatelet drugs.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Aspirin — See arm/group descriptions.
  Arms: DAPT group
Drug: Clopidogrel — See arm/group descriptions.
  Arms: DAPT group
Drug: Alteplase — See arm/group descriptions.
  Arms: IVT group

SUMMARY:
An open-label, blinded endpoint, randomized controlled trial that includes patients diagnosed with non-disabling, non-large vessel occlusion, acute minor stroke within 4.5 hours of onset. Eligible participants would be randomly assigned to the thrombolysis group (intravenous alteplase) and the dual antiplatelet group (oral aspirin plus clopidogrel). The primary outcome is the proportion of the excellent functional outcome (modified Rankin scale 0-1) at 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-80 years.
2. Diagnosed with acute ischemic stroke, NIHSS ≤ 5 and single item score ≤ 1 for vision, language, single limb, and no impairment of consciousness.
3. Time from symptoms onset to randomization within 4.5 hours; the onset time refers to the "Last Known Normal" (LKN).
4. Absence of large vessel occlusion on CTA.
5. Pre-stroke mRS ≤ 1.
6. Signed informed consent.

Exclusion Criteria:

1. Clinically confirmed valvular or non-valvular atrial fibrillation requiring anticoagulation therapy.
2. Intracranial hemorrhage or subarachnoid hemorrhage suggested by CT scan.
3. Acute coronary syndrome suggested by Electrocardiogram.
4. History of gastrointestinal bleeding.
5. Planned sequential IVT or endovascular treatment.
6. History of allergy to aspirin, clopidogrel, and/or alteplase.
7. Systolic blood pressure exceeding 185 mmHg and/or diastolic blood pressure exceeding 110 mmHg despite antihypertensive treatment.
8. Blood glucose ≤ 2.7 mmol/L.
9. Epileptic seizures during a stroke attack.
10. Recent trauma (<15 days).
11. Recent intracranial or spinal cord surgery, head trauma, or stroke (<3 months).
12. History of intracranial hemorrhage, aneurysm, vascular malformation, or brain tumor.
13. Active visceral hemorrhage (<22 days).
14. History of anticoagulant use within 24 hours prior to onset.
15. Platelets <100,000, PTT > 40 seconds on heparin, or PT > 15 or INR > 1.7, or known bleeding disposition.
16. Anticipated life expectancy < 3 months.
17. Pregnant or lactating women.
18. Participation in other clinical trials.
19. Any condition that, in the judgment of the investigator, makes the patient unsuitable for this study or where this study may impose a significant risk to the patient (e.g., inability to understand and/or comply with study procedures and/or follow-up due to psychiatric disorders, cognitive or emotional impairment).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-1 | 90(±7) days
  The proportion of the modified Rankin Scale score (mRS) 0-1 at 90 days.

SECONDARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-1 | 7(±1) days
  The proportion of the modified Rankin Scale score (mRS) 0-1 at 7 days or discharge (whichever occurred first).
Early neurological deterioration | 7(±1) days
  The incidence of early neurological deterioration at 7 days.
Recurrent stroke | 90(±7) days
  The incidence of recurrent stroke at 90 days.

OTHER OUTCOMES:
SAFETY OUTCOME: Symptomatic intracranial hemorrhage | 24 (±12) hours
  Symptomatic intracranial hemorrhage within 36 hours (according to Heidelberg criteria)
SAFETY OUTCOME: Mortality | 90(±7) days
  Mortality at 90 days
SAFETY OUTCOME: Any intracranial hemorrhage | 24 (±12) hours
  Any intracranial hemorrhage within 36 hours (according to Heidelberg criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China